CLINICAL TRIAL: NCT01408823
Title: Pharmacokinetics of Epsilon-Aminocaproic Acid in Children and Adolescents With Scoliosis Undergoing Posterior Spinal Fusion
Brief Title: Pharmacokinetics of Aminocaproic Acid in Scoliosis Surgery
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Children's Anesthesiology Associates, Ltd. (Other)
Responsible Party: Sponsor
Other Study IDs: 11-008205
Record Dates: First submitted 2011-07-13; First posted 2011-08-03 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-08

CONDITIONS: Scoliosis
Keywords: Pediatrics; Scoliosis; Pharmacokinetics; Hemorrhage; Orthopedic Surgery
MeSH Terms: conditions — Scoliosis; Hemorrhage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Idiopathic Scoliosis
- Non-idiopathic Scoliosis

SUMMARY:
This study will evaluate the pharmacokinetics of antifibrinolytic drug epsilon-aminocaproic acid (EACA) in children undergoing Posterior spinal fusion surgery (PSF) at The Children's Hospital of Philadelphia (CHOP) who receive EACA at the standard dose reported in the literature for this population and currently in use at CHOP.

DETAILED DESCRIPTION:
Posterior spinal fusion surgery (PSF) can be associated with significant blood loss, and perioperative transfusion is common. Various strategies have been employed to decrease intraoperative blood loss and reduce transfusion in children undergoing PSF. The intraoperative administration of the antifibrinolytic drug epsilon-aminocaproic acid (EACA) is one such strategy that has been shown to be effective in this regard. This study will evaluate the pharmacokinetics of EACA in children undergoing PSF at CHOP who receive EACA at the standard dose reported in the literature for this population and currently in use at CHOP.

ELIGIBILITY:
Inclusion Criteria:

1)Males or females age 8 to 18 years 2)Subjects undergoing posterior spinal fusion surgery 3)Subjects in whom aminocaproic acid administration is planned by the anesthesiology team 4)Parental/guardian permission (written informed consent) and when appropriate, child assent.

-

Exclusion Criteria:

1. Wards of the State are not eligible
2. Subjects with a history of abnormal renal function -

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and Adolescents scheduled to have posterior spinal fusion surgery at The Children's Hospital of Philadelphia
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2011-07; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters of EACA in participants undergoing Posterior Spinal Fusion | up to 15 hours
  The primary endpoint is the clearance of EACA

SECONDARY OUTCOMES:
Determine population-specific EACA dosing strategies based on the observed EACA pharmacokinetics | one year
  Population-specific EACA dosing strategies for patients with non-idiopathic and idiopathic scoliosis
Pharmacokinetic parameters of EACA in participants undergoing Posterior Spinal Fusion | up to 15 hours
  A secondary endpoint is the calculation of mean concentration levels of EACA in the body (AUC0-∞)
Pharmacokinetic parameters of EACA in participants undergoing Posterior Spinal Fusion | up to 15 hours
  A secondary endpoint is the clearance of EACA
Pharmacokinetic parameters of EACA in participants undergoing Posterior Spinal Fusion | up to 15 hours
  A secondary endpoint is the half-life of EACA
Pharmacokinetic parameters of EACA in participants undergoing Posterior Spinal Fusion | up to 15 hours
  A secondary endpoint is the volume of distribution of EACA

CONTACTS AND LOCATIONS:
Overall Officials: Paul Stricker, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Stricker PA, Gastonguay MR, Singh D, Fiadjoe JE, Sussman EM, Pruitt EY, Goebel TK, Zuppa AF. Population pharmacokinetics of ϵ-aminocaproic acid in adolescents undergoing posterior spinal fusion surgery. Br J Anaesth. 2015 Apr;114(4):689-99. doi: 10.1093/bja/aeu459. Epub 2015 Jan 13. PMID 25586726